CLINICAL TRIAL: NCT01943448
Title: Macular Hemorrhage in Myopic Eyes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201303121RINC
Record Dates: First submitted 2013-09-12; First posted 2013-09-17 (Estimated); Last update posted 2014-04-15 (Estimated); Status verified 2014-04

CONDITIONS: Macula Lutea Hemorrhage; High Myopia
Keywords: Macula Lutea Hemorrhage; High Myopia; Optical Coherence Tomography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
Visual impairment in high myopic eyes is mainly due to the different types of myopic maculopathies, such as diffuse or patchy atrophy, lacquer cracks and choroidal neovascularization. Macular hemorrhage was one of those complications. Despite choroidal neovascularization, simple hemorrhage from rupture of Bruch's membrane and choroidal microcirculation is also the cause of hemorrhage. The prognosis of those eyes with simple hemorrhage is generally good. However, some patients had persistently poor vision after the absorption of the hemorrhage. In the literature, the visual prognosis in those patients was reported to be associated with the microstructure change under the optical coherent tomography (OCT) or the presentation of the autofluorescence. The investigators will collect the patients with high myopia and presenting with macular hemorrhage. High resolution OCT and autofluorescence imaging will be used to analyze the change of the microstructure of retina and its correlation with the visual prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Myopia more than -6D
* Macular hemorrhage inside arcade
* Patients who are willing to visit our clinic and receive examination regularly for at least 1 year

Exclusion Criteria:

* Patients who cannot cooperate.
* Macular hemorrhage unrelated to myopia

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Myopia more than -6D
  2. Macular hemorrhage inside arcade
  3. Patients who are willing to visit our clinic and receive examination regularly for at least 1 year
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2013-08; Primary Completion 2015-05 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
visual acuity | 1 year
  visual acuity during follow up and its correlation to other factors

SECONDARY OUTCOMES:
Optical coherence tomography | 1 year
  Change of microstructure of the retina and choroid on OCT during follow up

CONTACTS AND LOCATIONS:
Overall Officials: Tzyy-Chang Ho, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- Department of Ophthalmology, National Taiwan University Hospital, Taipei, Taiwan